CLINICAL TRIAL: NCT07094906
Title: Neural and Vascular Modulation With Isometric Handgrip Training in Chronic Kidney Disease
Brief Title: Handgrip Exercise Training and CKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Jeanie Park, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00009157
Record Dates: First submitted 2025-07-25; First posted 2025-07-31 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Kidney Diseases
Keywords: Handgrip; Isometric handgrip exercise training (IHT); Blood pressure variability
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Isometric Handgrip Training (Experimental): The intervention is an 8-week isometric handgrip training protocol that consists of handgrip exercises performed by the participant at home, with a frequency of three sessions per week. Participants will log their exercise times as well as their perceived rate of exertion and recovery status throughout the 8 weeks.
  Interventions: Device: Isometric handgrip exercise training
- Sham Training (Sham Comparator): The intervention is an 8-week sham training protocol that consists of handgrip exercises performed by the participant at home, with a frequency of three sessions per week.
  Participants will log their exercise times as well as recovery status and training loads (borg scale) throughout the 8 weeks of intervention.
  Interventions: Device: Sham Training

INTERVENTIONS:
Device: Isometric handgrip exercise training — Maximum voluntary contraction (MVC) will be assessed first in both hands using a hand dynamometer with a digital display (Handexer HFEH20); the participant squeezes the hand dynamometer as hard as they can for 3 to 5 attempts to obtain the MVC. The intervention is an 8- week training protocol that consists of handgrip exercises performed by the participant at home. Each cycle of sustained handgrip exercise consists of sustained squeezing of the hand dynamometer at 30% of MVC for 2 minutes (i.e. isometric) followed by 1 minute of rest.
  Other Names: IHT
  Arms: Isometric Handgrip Training
Device: Sham Training — Each cycle of sustained handgrip exercise consists of sustained squeezing of the hand dynamometer at 3 - 5% of MVC rather than 30%.
  Arms: Sham Training

SUMMARY:
The purpose of this study is to find out if regular handgrip exercise performed at home can improve blood pressure at rest and during exercise in patients with chronic kidney disease (CKD).

This study is also intended to understand what causes an increase in blood pressure at rest and during exercise (i.e., increased adrenaline levels, or decreased ability of blood vessels to dilate). Patients with CKD will be recruited from primary care, Nephrology and other subspecialty Clinics throughout the Emory Healthcare System. Participants will attend 4 visits of 2-3 hours and 3 visits of 1-2 hours. The home exercise training will last for 8 weeks.

DETAILED DESCRIPTION:
The goal of this study is to learn more about if exercising the grip strength at home can improve blood pressure control. Patients with Chronic Kidney Disease (CKD) have a much higher risk of cardiovascular problems than healthy people. Early results show that patients with CKD have issues controlling their blood pressure. The investigators think that this type of exercise, where you use a grip device to squeeze, might help improve health by lowering blood pressure. Even though the American Heart Association recommends this kind of exercise, not many people are using it. The study population will consist of 50 patients with CKD in stages III and IV. They will do the grip exercise three times a week at home, squeezing a grip device four times for 2 minutes with each hand. The research team will also check their flight-or-flight control and artery health to see how this exercise training might help. The investigators will collect some blood samples to understand what changes are happening in their bodies. Patients with CKD will attend 4 visits of 2-3 hours and 3 visits of 1-2 hours. The home exercise training will last for 8 weeks. Therefore, the approximate study duration is around 12 weeks. Patients with CKD will be recruited from primary care, Nephrology and other subspecialty Clinics throughout the Emory Healthcare System. No bank for specimens or data will be maintained. The informed consent process will occur in-person. This study will help to find new ways to improve CKD cardiovascular health.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD (Stages IIIa and IV),
* Ages 45-85 years who do not regularly exercise (defined as exercising less than 20 minutes twice per week), willing and able to cooperate with the protocol.
* CKD Stages III and IV will be defined as reduction in estimated glomerular filtration rate (eGFR) to 15-59 cc/minute as calculated by the modified CKD-EPI equations.
* Patients with CKD must have stable renal function (no greater than a 20% reduction in eGFR over the prior 3 months).

Exclusion Criteria:

* Severe CKD (eGFR<15 cc/minute)
* Metabolic alkalosis (serum bicarbonate > 28 meq/L)
* Ongoing drug or alcohol abuse
* Diabetic neuropathy
* Any serious systemic disease that might influence survival
* Severe anemia with hgb level <10 g/dL
* Clinical evidence of congestive heart failure or ejection fraction below 35%, symptomatic heart disease determined by prior electrocardiogram, stress test, and/or history, treatment with central alpha agonists (clonidine)
* Uncontrolled hypertension with BP greater than 170/100 mm Hg
* Low blood pressure with BP less than 100/50
* Pregnancy or plans to become pregnant
* Current treatment with MAO inhibitors
* Inability to perform handgrip exercise

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in resting blood pressure (BP) | Baseline, 8-weeks post-intervention
  Resting BP will be recorded
Change in standard deviation BP variability | Baseline, 8-weeks post-intervention
  Resting beat-to-beat BP will be continuously measured for 10 min. Then, the standard deviation, and BP variability in mmHg will be calculated
Change in average real BP variability | Baseline, 8-weeks post-intervention
  Resting beat-to-beat BP will be continuously measured for 10 min. Then, the average variability in mmHg will be calculated.
Change in the coefficient of variation of BP variability | Baseline, 8-weeks post-intervention
  Resting beat-to-beat BP will be continuously measured for 10 min. Then, the coefficient of variation of BP variability in % will be calculated.
Change in Brachial artery flow-mediated dilation (FMD) | Baseline, 8-weeks post-intervention
  FMD of the brachial artery will be measured using doppler ultrasound. The image of the brachial artery will be obtained in the distal third of the arm (2-10 cm above the antecubital fossa) using a multi-frequency linear probe attached to a high-resolution Doppler US.
Change in Vascular stiffness | Baseline, 8-weeks post-intervention
  Vascular stiffness will be quantified as pulse wave velocity using applanation tonometry with a high-fidelity micromanometer. It will be reported in meters per second (m/s).

SECONDARY OUTCOMES:
Change in 24-hour ambulatory BP monitoring (ABPM) | Baseline, 8-weeks post-intervention
  ABPM will be performed with SpaceLab "On Trak" ambulatory BP monitors. Upper arm readings will be taken for at least 24 hours. BP measurements will be made every 20 minutes from 7 AM to 11 PM (daytime period) and every 30 minutes from 11 PM to 7 AM (nighttime period). Average BP in mmHg will be recorded.
Change in resting muscle sympathetic nerve activity (MSNA) | Baseline, 8-weeks post-intervention
  The tungsten microelectrode will be inserted under ultrasound guidance into the peroneal nerve to measure MSNA. Nerve signals are preamplified (gain 1000), amplified (gain 50-100), filtered (700-2000 Hz), rectified, and integrated (time constant 0.1 sec) to obtain a mean voltage display of sympathetic nerve activity that is recorded. Muscle sympathetic bursts are identified by visual inspection and expressed as burst frequency (bursts min).
Change in BP reactivity to cold pressor test (CPT) | Baseline, 8-weeks post-intervention
  The CPT will be performed by submerging the participant's hand in cold water (~0-4°C) up to the wrist for 1 minute. BP reactivity to the CPT in mmHg will be recorded.
Change in heart rate reactivity to cold pressor test (CPT) | Baseline, 8-weeks post-intervention
  Heart rate reactivity to the CPT in beats per minute will be recorded.
Change in MSNA reactivity to cold pressor test (CPT) | Baseline, 8-weeks post-intervention
  The MSNA reactivity in bursts/min will be recorded during the CPT using the tungsten microelectrode.
Change in BP reactivity to handgrip exercise | Baseline, 8-weeks post-intervention
  BP reactivity (in mmHg) to handgrip exercise, an isometric hand contraction at 30% of their maximal voluntary contraction (MVC) for 3 minutes followed by inflation of the BP cuff in their upper arm for another 3 minutes, will be recorded.
Change in heart rate reactivity to handgrip exercise | Baseline, 8-weeks post-intervention
  Heart rate reactivity in beats per minute will be recorded during the handgrip exercise.
Change in MSNA reactivity to handgrip exercise | Baseline, 8-weeks post-intervention
  The MSNA reactivity in bursts/min will be recorded during the handgrip exercise.
Change in skeletal muscle oxygenation during handgrip exercise | Baseline, 8-weeks post-intervention
  Skeletal muscle oxygenation will be calculated during handgrip exercise using Near-infrared spectroscopy (NIRS).
  NIRS will measure changes in oxyhemoglobin (oxygenated hemoglobin), deoxyhemoglobin (deoxygenated hemoglobin), and total hemoglobin. Percentage of oxyhemoglobin will be reported.
Change in interstitial muscle pH during handgrip exercise | Baseline, 8-weeks post-intervention
  Change in interstitial muscle pH during handgrip exercise will be assessed using NIRS.
Change in cardiac baroreflex sensitivity | Baseline, 8-weeks post-intervention
  The spontaneous cardiac baroreflex sensitivity expressed in milliseconds per mmHg (ms/mmHg) will be calculated at baseline, and at the end of the 8-week trial period.
Change in sympathetic baroreflex sensitivity | Baseline, 8-weeks post-intervention
  The spontaneous sympathetic baroreflex sensitivity expressed in bursts per 100 heartbeats per mmHg will be calculated at baseline, and at the end of the 8-week trial period.
Change in Inflammatory markers: C-Reactive Protein (CRP) | Baseline, 8-weeks post-intervention
  Blood will be collected at baseline, and at the end of the 8-week trial period to measure CRP.
Change in Inflammatory markers: Interleukin-6 (IL-6) | Baseline, 8-weeks post-intervention
  Blood will be collected at baseline, and at the end of the 8-week trial period to measure IL-6.
Change in Inflammatory markers: endothelin | Baseline, 8-weeks post-intervention
  Blood will be collected at baseline, and at the end of the 8-week trial period to measure endothelin.
Change in Inflammatory markers: asymmetric dimethyl arginine (ADMA) | Baseline, 8-weeks post-intervention
  Blood will be collected at baseline, and at the end of the 8-week trial period to measure ADMA.
Change in Inflammatory markers: phospholipase A2 (PLA-2) | Baseline, 8-weeks post-intervention
  Blood will be collected at baseline, and at the end of the 8-week trial period to measure PLA-2.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanie Park, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in this article after deidentification (text, tables, figures, and appendices) will be shared with investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be given upon request.